CLINICAL TRIAL: NCT04417231
Title: Selective Depletion of C-reactive Protein by Therapeutic Apheresis (CRP-apheresis) in Ischemic Stroke
Brief Title: CASTRO1 - Study on CRP Apheresis After Ischemic Stroke
Acronym: CASTRO1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sufficient recruitment of study patients based on the existing (and repeatedly adjusted) inclusion and exclusion criteria is not possible within a reasonable period of time
Sponsor: Pentracor GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-05 CASTRO1
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-01

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apheresis group (Experimental): 10 patients receive a maximum of 3 apheresis treatments at intervals of 24 ± 12 hours each (from the beginning of the preceding treatment). The first treatment starts within 72 hours after infarction or, in case of an unclear time window, within presumed 72 hours after the patient was last seen free of symptoms. No further treatments are carried out if the CRP concentration before the start of a treatment is <10 mg/l or if the patient has been discharged from hospital.
  For each treatment, 1.5 - 2.5 times the plasma volume is processed. The duration of each treatment is approximately 4-6 hours.
  Interventions: Device: CRP apheresis
- Control group (No Intervention): 10 patients of the control group receive the same examinations as arm 1 (verum group) but no apheresis treatments after ischemic stroke.

INTERVENTIONS:
Device: CRP apheresis — Selective CRP apheresis by use of the "PentraSorb"-CRP
  Arms: Apheresis group

SUMMARY:
CASTRO1 is a study to investigate the reduction of C-reactive protein (CRP) by therapeutic apheresis (CRP-apheresis) in patients after primary treatment of ischemic stroke.

The term therapeutic apheresis commonly refers to medical procedures, where pathogenic constituents are being removed from the circulating blood. Elimination is performed by adsorbers outside the body in an extracorporeal circulation. For removal of the pathogenic substances the plasma is separated from the blood (circulation) to pass the adsorber. The purified plasma is merged with the solid blood components thereafter and returned to the patient.

The adsorber "PentraSorb® CRP" used for CRP apheresis is CE-certified. It is designated to the selective depletion of C-reactive protein from human blood.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and efficacy of CRP apheresis in patients following ischemic stroke. CRP apheresis is to be conducted with the aim of reducing cerebral damage following the guideline-appropriate primary therapy of ischemic stroke.

A possible protective effect of CRP apheresis will be assessed by clinical scores, laboratory determination of immunologic parameters and determination of the size of the infarct area by magnetic resonance imaging (MRI).

The study will be randomized, controlled and monocentric.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic stroke with determination of infarct size by imaging (MRI)
* NIHSS 1-24
* CRP increase ≥ 5 mg/l within presumed 72 hours after stroke and/or CRP value > 10 mg/l
* written informed consent of the patient or his legal representative

Exclusion Criteria:

* age < 18 years
* Severe dysphagia (danger of aspiration pneumonia)
* Clinical or laboratory evidence of a severe systemic infection
* Participation in other interventional studies
* Contraindications against apheresis therapy
* Modified Rankin Scale (mRS) before index event ≥ 3
* Intracranial hemorrhage
* Epileptic seizure in the context of the acute event
* Pregnancy, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of CRP apheresis | 24 hours after each apheresis
  Incidence of expected and unexpected adverse effects

SECONDARY OUTCOMES:
Stroke Severity | before first apheresis and 6 ± 3 days after infarction and 12 ± 2 weeks after infarction
  National Institute of Health Stroke Scale (NIHSS) score - ranging from 0-42 - higher values represent a worse outcome
Functional Outcome | before first apheresis and 6 ± 3 days after infarction and 12 ± 2 weeks after infarction
  Modified ranking scale (mRS) score - ranging from 0-6 with higher scores signifying worse outcome
Dependency | 6 ± 3 days after infarction and 12 ± 2 weeks after infarction
  Barthel Index (BI) - ranging from 0-100 with higher scores signifying better outcome
Infarct size | 6 ± 3 days after infarction and 12 ± 2 weeks after infarction
  Infarct growth measured via diffusion-weighted imaging (DWI)-FLAIR volume change
Concentration of inflammatory biomarkers (CRP, IL-6, SAA) | 0-7 days after infarction
  CRP, Interleukin-6, and serum amyloid A are determined twice daily until discharge of the patient (for a maximum of 7 days).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Dorst, PD Dr. med., Principal Investigator — Universitätsklinik Ulm, Abteilung für Neurologie
Locations (1):
- Abteilung für Neurologie, Universität Ulm, Ulm, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No